CLINICAL TRIAL: NCT02586727
Title: Role of Intravitreal Aflibercept Injection for the Treatment of Radiation Maculopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCH-1-012015
Record Dates: First submitted 2015-08-20; First posted 2015-10-26 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Adverse Effect of Radiation Therapy
Keywords: Radiation Retinopathy; aflibercept
MeSH Terms: conditions — Radiation Injuries | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- six week dosing regimen arm (Active Comparator): Patients will receive an intravitreal aflibercept injection the first visit, and then again every six weeks. Treatment will be given at each visit.
  Interventions: Drug: aflibercept
- treat and extend dosing regimen arm (Active Comparator): Patients will receive an intravitreal aflibercept injection the first visit, again at the second visit at 6 weeks, and then begin treat and extend from second injection forward. Patients with decreased radiation maculopathy by one grade or more will extend re-evaluation by two weeks. Patients with increased radiation maculopathy by one grade or more will have re-evaluation decreased by one week. Patients that show no maculopathy grade change will remain at the same re-evaluation interval.
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — This study will consist of 2 simultaneous treatment arms of aflibercept: A six week dosing regimen arm and a treat and extend (TAE) dosing regimen arm, total duration 54 weeks. In the TAE arm the patients will receive an intravitreal aflibercept injection first visit, again at the second visit at 6 weeks, and then begin treat and extend from second injection forward.
  Other Names: Eylea

SUMMARY:
The primary objective of the study is to assess the safety of intravitreal aflibercept injection in treating visually compromising radiation maculopathy secondary to treatment of uveal melanoma by iodione-125 brachytherapy. The study will consist of two arms of 25 patients each (totaling 50 patients). Subjects in arm 1 will undergo treatment every 6 weeks. Subjects in arm 2 will undergo treatment and if improvement is documented at the following evaluation the next treatment will be extended by two weeks. Secondary objectives of the study include evaluation and analysis of visual acuity, number of injections, macular edema, and vascular activity between both arms.

DETAILED DESCRIPTION:
This study will consist of 2 simultaneous treatment arms: A six week dosing regimen arm and a treat and extend (TAE) dosing regimen arm, total duration 54 weeks. In the TAE arm the patients will receive an intravitreal aflibercept injection first visit, again at the second visit at 6 weeks, and then begin treat and extend from second injection forward. Treatment will be given at each visit. Patients with improved radiation maculopathy (SD-OCT analysis) will extend re-evaluation by two weeks (e.g. first interval 6 weeks; second interval 10 weeks; third interval 12 weeks, etc). Patients with increased radiation maculopathy (SD-OCT analysis) will have re-evaluation decreased by one week. Both arms will consist of 25 subjects (eyes). Fluorescein angiography will be completed at baseline, after the 4th injection (or within three weeks of week 24 for the TAE arm), and at the end of the study in all patients. Spectral domain OCT, and clinical evaluation including visual acuity will be assessed every visit in all patients. Radiation maculopathy will be graded every visit in all patients in a blinded fashion using the following classification system: Grade 1 indicates extrafoveal, noncystoid edema; grade 2, extrafoveal cystoid edema; grade 3, foveal noncystoid edema; grade 4, mild-to-moderate foveal cystoid edema; grade 5, severe foveal cystoid edema and grade 6 subretinal fluid. All patients will undergo comprehensive evaluation including adverse event questioning at each study timepoint. Patients in the six-week dosing arm will receive a total of 9 intravitreal aflibercept injections during the study window while the TAE treatment group will receive a maximum of 9 with a minimum of 5.

ELIGIBILITY:
Inclusion Criteria:

* A Patient must meet the following criteria to be eligible for inclusion in the study:

  1. 21 years of age and over
  2. 20/800 or better visual acuity
  3. Must have received previous treatment for radiation maculopathy within the last 4-26 weeks
  4. Any presence of macular edema (evaluated by SD-OCT) caused by radiation retinopathy
  5. Willing and able to comply with clinic visits and study-related procedures
  6. Provide signed informed consent

Exclusion Criteria:

* A patient who meets any of the following criteria will be excluded from the study:

  1. Patients less than 21 years of age.
  2. Patients with mental disability or any other condition that precludes the acquisition of an sdOCT image such as (nystagmus, neck disease, etc.)
  3. Patients who have previously been treated with intravitreal triamcinolone acetonide for macular edema (signs of recalcitrant disease)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy G Murray, MD, MBA, Principal Investigator — Murray Ocular Oncology & Retina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Six Week Dosing Regimen Arm | Treat and Extend Dosing Regimen Arm
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Six Week Dosing Regimen Arm | Treat and Extend Dosing Regimen Arm | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 8 | 13 | 21
Age, Continuous [Mean (Full Range); unit: Years] | 62 [40 to 79] | 67.3 [40 to 81] | 64.7 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 8 | 12 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 19 | 18 | 37
  Hispanic | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Best Corrected Visual Acuity (BCVA) in Patients Treated With Intravitreal Aflibercept Injections for the Management of Radiation Maculopathy.
Description: BCVA will be measured with letter optotypes. A lower value indicates a better outcome.
Time Frame: 12 months
Population: Baseline study entry mean BCVA was 20/63 (Logmar 0.498)
Measure: Mean (Full Range); unit: Log MAR (Visual Acuity)
Arm/Group | Six Week Dosing Regimen Arm | Treat and Extend Dosing Regimen Arm
Number analyzed (Participants) | 20 | 20
Log MAR (Visual Acuity) | 0.425 [0 to 1.602] | 0.548 [0.097 to 1.602]

2. Secondary Outcome: Role of Intravitreal Aflibercept Injection on Central Retinal Thickness for the Treatment of Radiation Maculopathy.
Description: Central retinal thickness will be evaluated with OCT. A lower value considered a better outcome.
Time Frame: 12 months
Measure: Mean (Full Range); unit: microns
Units Other Than Participants: eye
Arm/Group | Six Week Dosing Regimen Arm | Treat and Extend Dosing Regimen Arm
Number analyzed (Participants) | 20 | 20
Number analyzed (eye) | 20 | 20
microns | 298 [154 to 482] | 294 [192 to 595]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Six Week Dosing Regimen Arm | Treat and Extend Dosing Regimen Arm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT02586727/Prot_SAP_000.pdf